CLINICAL TRIAL: NCT02859844
Title: Transcutaneous Tibial Nerve Stimulation for Treating Neurogenic Lower Urinary Tract Dysfunction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Termination after a few pilot participants due to further protocol development
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016-01016
Record Dates: First submitted 2016-06-30; First posted 2016-08-09 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Neurogenic Bladder Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- TTNS ON (Experimental): Transcutaneous tibial nerve stimulation
  Interventions: Device: Transcutaneous Tibial Nerve Stimulation (TTNS)
- TTNS OFF (Sham Comparator): Sham/placebo stimulation
  Interventions: Device: Transcutaneous Tibial Nerve Stimulation (TTNS)

INTERVENTIONS:
Device: Transcutaneous Tibial Nerve Stimulation (TTNS)

SUMMARY:
Many patients with neurological diseases suffer from neurogenic lower urinary tract dysfunction (NLUTD), which often severely impairs quality of life, due to urinary urgency with or without incontinence and voiding dysfunction. In addition, the upper urinary tract may be jeopardized because of high intravesical pressure caused by detrusor overactivity with concurrent detrusor-sphincter-dyssynergia and/or low bladder compliance. The treatment of NLUTD is a challenge since conventional conservative therapies often fail and more invasive treatments such as intradetrusor onabotulinumtoxinA injections, bladder augmentation and urinary diversion have to be considered. Neuromodulation therapies including tibial nerve stimulation (TNS) may be alternative non-invasive treatment options. Indeed, TNS is an effective and safe treatment for idiopathic overactive bladder proven in randomized controlled trials (RCTs), but its value in neurological patients is unclear. In a recent systematic review, the investigators found evidence that TNS might become a promising treatment option for NLUTD, however, more reliable data from well-designed RCTs are urgently needed to reach definitive conclusions. However, the investigators study will be the first adequately sampled and powered, randomized, placebo-controlled, double-blind trial assessing transcutaneous TNS (TTNS) for NLUTD. This trial will provide significant insights into the efficacy of TTNS in patients suffering from NLUTD and in the case that this treatment is really effective in the neurological population, the investigators findings would completely revolutionize the management of NLUTD in daily clinical practice. Moreover, this interdisciplinary trial will relevantly influence the neurological and urological approach in the management of NLUTD promoting future collaborative projects improving patients' medical care and underlying the pioneering role of Switzerland in the rapidly developing and ambitious research field of neuro-urology.

ELIGIBILITY:
Inclusion Criteria:

* Refractory LUTD due to a neurological disorder:
* Urgency frequency syndrome and/or urgency incontinence refractory to antimuscarinics (pharmacotherapy for at least 4 weeks with at least 2 antimuscarinics)
* Chronic urinary retention refractory to alpha-blocker (pharmacotherapy with an alpha-blocker for at least 4 weeks)
* Combination of urgency frequency syndrome and/or urgency incontinence and chronic urinary retention refractory to antimuscarinics (pharmacotherapy for at least 4 weeks with at least 2 antimuscarinics) and alpha-blocker (pharmacotherapy with an alpha-blocker for at least 4 weeks)
* Age >18 years
* Informed consent

Exclusion Criteria:

* Botulinum A toxin injections in the detrusor and/or urethral sphincter in the last 6 months
* Age <18 years
* Pregnancy
* Individuals especially in need of protection (according to Research with Human Subjects published by the Swiss Academy of Medical Sciences www.samw.ch/en/News/News.html)
* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-10; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Number of voids | 6 weeks
Number of leakages | 6 weeks
Number of used pads | 6 weeks
Post void residual (mL) | 6 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - EOC-Ospedale regional Bellinzona e Valli, Bellinzona
  - Universitätsklinik Balgrist, Zurich